CLINICAL TRIAL: NCT02613611
Title: Screening for Human Papilloma Virus in Urine and Pap Smear.A Comparative Study.
Brief Title: HPV Screening (Human Papilloma Virus)
Acronym: HPV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, suzy abdelaziz Abdelhamid, lecturer of obgyn., Kasr El Aini Hospital
Other Study IDs: Obgyn.. .. ..
Record Dates: First submitted 2015-11-21; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: HPV Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Examination of cervical &urine samples for HPV

DETAILED DESCRIPTION:
500 females attending colposcopy kasrelaini unit are included. History including age and parity is taken.urine samples are taken. Colposcopy will be done. Pap smear will be taken and sent for pathology.

ELIGIBILITY:
Inclusion Criteria:

* all females attending colposcopy kasrelaini unit aging 18_45 years

Exclusion Criteria:

* females with known cervical cancer
* females less than 18 or more than 45

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 500 females attending colposcopy kasrelaini unit aging 18_45 years
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive urine test for HPV Number of patients with positive pap smear. | 3 months